CLINICAL TRIAL: NCT04864353
Title: A Guided Internet-delivered Intervention for Adults With Residual Cognitive Symptoms After Major Depressive Disorder: Study Protocol for a Randomized Controlled Trial Investigating Clinical Effects
Brief Title: Internet-delivered Intervention Targeting Residual Cognitive Symptoms After Major Depressive Disorder
Acronym: RestDep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 204287
Record Dates: First submitted 2021-04-21; First posted 2021-04-28 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Cognitive Remediation; Cognitive Impairment; Major Depression in Remission
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Masking Description: The assessor do not allocate the participant to the intervention or waitlist group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention (Experimental): Participants will after baseline receive a guided intervention with weekly therapist support.
  Interventions: Behavioral: RestDep: Internet-delivered intervention targeting residual cognitive symptoms
- Control: Waitlist (No Intervention): Participants will not receive intervention until 7 weeks after baseline.

INTERVENTIONS:
Behavioral: RestDep: Internet-delivered intervention targeting residual cognitive symptoms — The intervention is fully digital with weekly telephone guidance. Key intervention elements are 1) psychoeducation, 2) attention training, 3) strategy training. Cognitive domains as attention, memory and executive functions are covered and rumination.
  Arms: Experimental: Intervention

SUMMARY:
Background: Cognitive impairment and difficulties are frequently observed in individuals suffering from major depressive disorder. These impairments and difficulties can persist into remission as residual cognitive symptoms. Consequently affecting daily life functioning and quality of life for those affected. Few scalable interventions have targeted these symptoms and measured long-term clinical effects such as depression relapse.

DETAILED DESCRIPTION:
Background:Cognitive impairment and difficulties are frequently observed in individuals suffering from major depressive disorder. These impairments and difficulties can persist into remission as residual cognitive symptoms. Consequently affecting daily life functioning and quality of life for those affected. Few scalable interventions have targeted these symptoms and measured long-term clinical effects such as depression relapse.

Objectives: The aim is to assess the clinical effects of an intervention targeting residual cognitive symptoms after major depressive disorder. More specifically, if residual cognitive symptoms would be significantly decreased from pre- to post-treatment and remain stable at the 6-month and 2 year follow-up.

Methods: the study is a randomized, waitlist controlled trial including a total of 60 participants (30 in each arm). Primary measures are residual cognitive symptoms measured by the Behavioral Rating Inventory of Executive Functions Adults (BRIEF-A) and Perceived Deficit Questionnaire 5 (PDQ-5). Secondary outcome measures are Depression measured by Montgomery Aasberg Depression Rating Scale and Patient Health Questionnaire 9 and 2 (PHQ-9 and PHQ2), Satisfaction with life measured by Satisfaction with life scale (SWLS), Credibility measured by the Treatment Credibility and Expectation Scale, Rumination measured by the Rumination Response Scale (RRS), Depression screening assessed using the MINI International Psychiatric Interview, Usage data measured by number of log-ins, session length and days in treatment. Quantitative statistical methods will be used to analyze data.

Discussion: The results from the study will contribute to field of internet interventions and provide former depressed adults with an easy access intervention in the treatment of residual cognitive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Previously received treatment for major depressive disorder in primary or secondary healthcare services
* Reporting a history of major depressive disorder symptoms assess using the MINI. few or minor depression symptomss (< 12 MADRS)
* Not meeting criteria for major depressive disorder measured by the MINI)
* Self-reporting residual cognitive symptoms that affects daily functioning (assessed by clinical psychologist)
* No changes in anti-depressant medication under the study period
* Age between 18 and 65 years
* Read and write Norwegian
* Internet and telephone access.

Exclusion Criteria:

* Self-reported substance abuse
* Neurological conditions or damage (e.g. autism, cerebral haemorrhage, and brain tumour)
* Bipolar disorder
* Psychosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Behaviour Rating Inventory Of Executive Function-Adult | 2.5 years
  The Behavior Rating Inventory of Executive Function-Adult (BRIEF-A; Roth, Isquith, & Gioia, 2005) is a 75-item self-report questionnaire designed to measure adults' behaviors associated with executive problems.
Perceived Deficit Questionnaire 5 | 2.5 years
  Brief assessment of subjective cognitive difficulties and covers problems with concentration (e.g. "trouble concentrating on things like watching a television program or reading a book?"), memory (e.g. "forget what you talked about after a telephone conversation?"), and executive functioning (e.g. "have trouble getting things organized?"). Every item is rated on a scale of 0 (Never) to 4 (Almost always) to yield a sum score of 0 to 20, with higher scores indicating greater severity of cognitive symptoms.

SECONDARY OUTCOMES:
Rumination Response Scale | 2.5 years
  The Rumination Response Scale (RRS; Treynor, Gonzalez, & Nolen-Hoeksema, 2003) is a questionnaire frequently used to assess rumination in depression. The 22-item RRS measures the current degree of ruminative responses to depressed mood.
Montgomery Aasberg Depression Rating Scale | 2.5 years
  The Montgomery Åsberg Depression Rating Scale Self-report (MADRS-S; Svanborg & Åsberg, 2001) is a self-report questionnaire measuring depressive symptoms during the past three days. The MADRS-S consists of 9 items where the following symptoms are rated on a seven-point scale ranging from 0 to 6.
Patient Health Questionaire 9 and 2 | 2.5 years
  The Patient Health Questionnaire-9 (PHQ-9: Kroenke et al., 2001) is a self-report tool used to assess the presence and severity of depressive symptoms. Reliability and validity of the tool have indicated it has sound psychometric properties. Internal consistency of the PHQ-9 has been shown to be high.
The Satisfaction With Life Scale | 2.5 years
  The SWLS (Kobau et al., 2010) is a short 5-item instrument designed to measure global cognitive judgments of satisfaction with one's life. The scale usually requires only about one minute of a respondent's time.
The Credibility/Expectancy Questionnaire | 8 months
  The Credibility/Expectancy Questionnaire (Borkovec & Nau, 1972) measures treatment credibility and expectancy. Participants rated perceived treatment credibility and expectancy on a scale from 0 to 10 were higher scores indicated better treatment credibility or expectancy.
Log-ins | 8 months
  Number of sessions were participants have logged into the intervention during the intervention period.
Session length | 8 months.
  Average length of each log-in during the intervention period.
Days in treatment | 8 months
  Number of days in intervention from receiving intervention until completion.

CONTACTS AND LOCATIONS:
Overall Officials: Tine Nordgreen, PhD, Principal Investigator — Projectleader
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Myklebost SB, Heltne A, Hammar A, Nordgreen T. Efficacy of an internet-delivered cognitive enhancement intervention for subjective residual cognitive deficits in remitted major depressive disorder: A randomized crossover trial. J Affect Disord. 2024 Nov 1;364:87-95. doi: 10.1016/j.jad.2024.08.035. Epub 2024 Aug 12. PMID 39142571